CLINICAL TRIAL: NCT02205645
Title: A Prospective Open-Label Study to Evaluate the Safety of the Meniscal Repair Scaffold, FibroFix™ Meniscus, in the Treatment of Meniscal Defects
Brief Title: Initial Safety Evaluation of FibroFix™ Meniscus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety. Devices explanted. 12m post-explant safety f/u as agreed with UK MHRA
Sponsor: Orthox Limited (Industry)
Collaborators: Avon Orthopaedic Centre, North Bristol NHS Trust, Bristol UK (Unknown); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORX/2014/FM01
Record Dates: First submitted 2014-07-23; First posted 2014-07-31 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2017-04

CONDITIONS: Other Tear of Medial Meniscus, Current Injury
Keywords: medial; meniscus; scaffold; repair; tear; injury
MeSH Terms: conditions — Lacerations; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FibroFix™ Meniscus scaffold (Experimental): The test article for this study is the FibroFix™ Meniscus scaffold, which has been developed for repair of defects of the meniscus. It is a silk derived product developed to functionally replace the excised unstable meniscus following a meniscal tear.
  Interventions: Device: FibroFix™ Meniscus scaffold

INTERVENTIONS:
Device: FibroFix™ Meniscus scaffold — The test article for this study is the FibroFix™ Meniscus scaffold supplied by Orthox Ltd. The FibroFix™ Meniscus scaffold has been developed for repair of defects of the meniscus.
  The FibroFix™ Meniscus scaffold used in this study is a silk derived product developed to functionally replace the excised unstable meniscus following a meniscal tear.

SUMMARY:
Initial evaluation of safety and performance of FibroFix™ Meniscus scaffold

DETAILED DESCRIPTION:
The safety of the FibroFix™ Meniscus scaffold will be evaluated in 10 patients scheduled for elective arthroscopic medial meniscus partial resection or treatment of asymptomatic medial meniscal defect

ELIGIBILITY:
Inclusion Criteria:

* The subject (or guardian, if appropriate) has signed and dated a specific informed consent form
* The subject is over the age of 18
* The subject is able to comply with the protocol-defined preoperative procedures, the postoperative clinical and radiographic evaluations and the recommended rehabilitation regimen as determined by the investigator
* The subject has a diagnosis of an MRI or arthroscopically confirmed irreparable medial meniscus defect
* The meniscal defect should represent 25% or more of the meniscus and be amenable to repair
* The peripheral meniscal rim must be present
* The subject has a functionally intact anterior cruciate ligament
* Haemoglobin >9g/dL and platelet count >100,000/mm3 prior to Day 1
* No contraindication to general anaesthetic
* Female subjects of child-bearing potential: a negative urine pregnancy test

Exclusion Criteria:

* The subject has a functionally deficient anterior cruciate ligament
* The subject has concomitant posterior cruciate ligament insufficiency of the involved knee or a concomitant injury that interferes with the subject's ability to comply with the recommended rehabilitation program
* The subject has a diagnosis of untreatable Grade IV Outerbridge Scale degenerative cartilage disease in the involved knee joint
* Patients demonstrating an active local or systemic infection
* Any condition, which in the judgment of the Investigator would preclude adequate evaluation of the FibroFix™ Meniscus scaffold and clinical outcome.
* The subject has a history of confirmed anaphylactoid reaction
* The subject has received local administration of any type of corticosteroid or systemic administration of antineoplastic, immunostimulating, or immunosuppressive agents within 180 days prior to the scheduled surgery
* The subject has evidence of osteonecrosis of the involved knee
* The subject has a medical history that includes a confirmed diagnosis of rheumatoid or inflammatory arthritis, or relapsing polychondritis
* If female and of child-bearing potential: evidence of a positive pregnancy test or a stated intention to become pregnant in the next 6-12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  Number of participants with Adverse Events

SECONDARY OUTCOMES:
Safety | 7 years
  Number of participants with Adverse Events
Functional assessment | 7 years
  Assessments will be made using recognized and validated tools: Tegner Index, Lysholm Score, International Knee Documentation Committee (IKDC) Score and range of motion of knee

OTHER OUTCOMES:
Pain scores | 12m
  Assessments will be made using recognized and validated tools: Tegner index, Lysholm score, International Knee Documentation Committee (IKDC) score, VAS scale
Functional assessment | 12m
  Assessments will be made using recognized and validated tools: Tegner Index, Lysholm Score, International Knee Documentation Committee (IKDC) score and range of motion of knee
Post operative infection | 12m
  Diagnosis of infection will be made on clinical grounds. If infection is diagnosed, a confirmatory bacterial culture will be collected and analysed locally. Assessment will include the patient, tissues around the wound and the wound itself.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Blom, Professor, Principal Investigator — University of Bristol
Locations (1):
- Southmead Hospital, Bristol, United Kingdom